CLINICAL TRIAL: NCT01303601
Title: Efficacy of Olanzapine Monotherapy for Treatment Bipolar Ⅰ Depression: a Randomized, Double-blind, Placebo Controlled Study
Brief Title: Efficacy of Olanzapine Monotherapy for Treatment Bipolar Ⅰ Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: China Medical University, China (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MWang
Record Dates: First submitted 2011-02-24; First posted 2011-02-25 (Estimated); Last update posted 2011-02-25 (Estimated); Status verified 2008-12

CONDITIONS: Bipolar Disorder; Depression, Bipolar
Keywords: Olanzapine; Monotherapy; bipolar Ⅰ depression
MeSH Terms: conditions — Bipolar Disorder | interventions — Olanzapine; Starch

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- olanzapine (Experimental)
  Interventions: Drug: olanzapine
- placebo (Placebo Comparator)
  Interventions: Drug: Starch

INTERVENTIONS:
Drug: olanzapine — Tablet The initial dose of olanzapine was 5mg daily and raised to 10 mg/day. After week 1, flexible dosing was allowed based on symptom response, up to 20 mg daily, as tolerated.
  daily 6 weeks
  Arms: olanzapine
Drug: Starch
  Arms: placebo

SUMMARY:
Olanzapine may have some antidepressant properties and olanzapine monotherapy has been shown efficacy in bipolar depressive episodes in retrospective studies. However, there has been no prospective study about the monotherapy of olanzapine. The investigators conducted a randomized, placebo-controlled study to test the efficacy of olanzapine monotherapy for treatment of the depressed phase of bipolar disorder.

DETAILED DESCRIPTION:
The study was designed as a double-blind randomized controlled trial, with research assessors and patients intended to be blind to the intervention status. The staff members performing the assessment were not involved in implementing any aspect of the intervention.68 patients were randomized to assigned 6 weeks by olanzapine or placebo. Medications were provided in double-blind fashion. The assessments include Montgomery-Asberg Depression Rating Scale, Young Mania Rating Scale, clinical Global Impressions-Severity of Illness scale, Clinical Global Impressions-Improvement scale, response and remission rates, and Treatment Emergent Symptom Scale.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with clinical diagnosis of bipolarⅠdisorder
* MADRS total score ≥ 20
* CGI-S rating ≥ 4
* Normal results of physical examinations, laboratory and electrocardiogram tests
* Being taken care of by a guardians during the trial

Exclusion Criteria:

* Pregnant or lactating women
* YMRS total score ≥ 15
* Treatment with olanzapine within 3 months prior to study entry
* Retrospective history of poor antidepressive response to or intolerance of olanzapine
* Mental retardation
* Addictive disorder
* Diabetes mellitus
* Dyslipidaemia
* Cardiovascular diseases
* Hypertension

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2009-01; Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale | once weekly

SECONDARY OUTCOMES:
The percentage of participants with a change in MADRS total score ≥50% from baseline as a measure of interventional response | once
The percentage of participants with an endpoint (last observation available) MADRS total score ≤12 as a measure of interventional remission | once
Young Mania Rating Scale | once weekly
Clinical Global Impressions-Severity of Illness Scale | once weekly
Clinical Global Impressions-Improvement Scale | once weekly

CONTACTS AND LOCATIONS:
Overall Officials: Man Wang, M.D., Study Director — First Hospital of China Medical University
Locations (1):
- Department of Psychiatry, the First Hospital of China Medical University, Shenyang, Liaoning, China